CLINICAL TRIAL: NCT03794908
Title: Bright Light Treatment at Home to Improve Symptom Management of Fibromyalgia Syndrome
Brief Title: Light Treatment to Improve Symptom Management of Fibromyalgia Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Principal Investigator, Helen Burgess, Professor of Psychiatry, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: HUM00151160; 1R21NR016930-01A1 (NIH)
Record Dates: First submitted 2019-01-03; First posted 2019-01-07 (Actual); Results first posted 2022-10-05 (Actual); Last update posted 2022-10-05 (Actual); Status verified 2022-09

CONDITIONS: Fibromyalgia; FMS
Keywords: Circadian timing; Pain; Light
MeSH Terms: conditions — Fibromyalgia; Pain

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: The outcome assessors and participants were blinded to condition. The PI and lab manager remained unblinded, and performed the fidelity and side-effects assessments. Participants were asked and reminded throughout the study to only speak about their light treatment with either the PI or lab manager.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Light therapy A (Bright) via the Re-Timer® (Experimental): * 60 minutes/day
  * For the first hour after waking
  Interventions: Device: Light therapy A (Bright) via the Re-Timer®
- Light therapy B (Dim) via the Re-Timer® (Active Comparator): * 60 minutes/day
  * For the first hour after waking
  Interventions: Device: Light therapy B (Dim) via the Re-Timer®

INTERVENTIONS:
Device: Light therapy A (Bright) via the Re-Timer® — Subjects will conduct light treatment in the mornings at home for one hour using Re-timer®.
  Other Names: Re-Timer®
  Arms: Light therapy A (Bright) via the Re-Timer®
Device: Light therapy B (Dim) via the Re-Timer® — Subjects will conduct light treatment in the mornings at home for one hour using Re-timer®.
  Other Names: Re-Timer®
  Arms: Light therapy B (Dim) via the Re-Timer®

SUMMARY:
The purpose of this study is to determine the effect a morning light treatment has on improving physical function, pain intensity, and pain sensitivity in people with fibromyalgia syndrome (FMS).

ELIGIBILITY:
Inclusion Criteria:

• Meet criteria for Fibromyalgia syndrome (FMS)

Exclusion Criteria:

* Significant chronic disease
* Severe hearing or memory problems
* Pending medical leave applications at workplace
* Current pregnancy, breastfeeding, or actively trying to get pregnant
* Night work or travel outside the eastern time zone within 1 month of the study
* Other research participation
* Frequent number of special events during study period (weddings, concerts, exams, etc).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2019-01-31 (Actual); Primary Completion 2021-07-15 (Actual); Study Completion 2021-07-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Helen Burgess, Principal Investigator — University of Michigan
Locations (1):
- The University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: Yes
The researchers are open to sharing data by any appropriate mechanism indicated by NIH program staff.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: After scientific papers are accepted for publication and the data will be available for 7 years after study completion.
Access Criteria: Researchers requesting data will first have to sign a data sharing agreement, agreeing to the conditions of use governing access to the public release data, including restrictions against attempting to identify study participants, electronically securing the data while in use, destruction of the data after analyses are completed, reporting responsibilities, restrictions on redistribution of the data to third parties, no use of the data for commercial purposes and proper acknowledgement of the data resource.

REFERENCES:
- See also: Additional study information and application to apply for study — https://is.gd/Fibrolight

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 60 participants were enrolled, and 57 participants were randomized.
Groups:
- Light Therapy A (Bright) Via the Re-Timer®: * 60 minutes/day
  * For the first hour after waking
  Light therapy A (bright light) via the Re-Timer®: Subjects conducted light treatment in the mornings at home for one hour using Re-timer®.
- Light Therapy B (Dim) Via the Re-Timer®: * 60 minutes/day
  * For the first hour after waking
  Light therapy B (dim light) via the Re-Timer®: Subjects conducted light treatment in the mornings at home for one hour using Re-timer®.
Period: Overall Study
Arm/Group | Light Therapy A (Bright) Via the Re-Timer® | Light Therapy B (Dim) Via the Re-Timer®
Started | 29 | 28
Began Use of Re-Timer | 27 | 27
Completed | 27 | 27
Not Completed | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Light Therapy A (Bright) Via the Re-Timer® | Light Therapy B (Dim) Via the Re-Timer® | Total
Number analyzed (Participants) | 29 | 28 | 57
Age, Continuous [Mean (Standard Deviation); unit: Years] | 41.3 (13.7) | 42.4 (13.1) | 41.8 (13.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 | 27 | 55
  Male | 1 | 1 | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 0 | 3
  Not Hispanic or Latino | 26 | 28 | 54
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 3 | 4
  White | 26 | 22 | 48
  More than one race | 0 | 2 | 2
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 29 | 28 | 57
Apnea-Hypopnea Index [Mean (Standard Deviation); unit: Events per hour] — Number of pauses in breath per hour during nighttime sleep. Population: Participants who elected not to wear the watchPAT device were not included in the analysis.
  Events per hour
    number analyzed (Participants) | 29 | 25 | 54
    (all) | 16.33 (14.3) | 11.2 (10.2) | 14.0 (12.7)

OUTCOME MEASURES:

1. Primary Outcome: Fibromyalgia Impact Questionnaire, Revised (FIQ-R) Score
Description: The FIQR consisted of 21 questions. Each question had 11 boxes similar to a visual analog scale. Questions covered the difficulty associated with various physical activities and the severity of symptoms. The score for the questions was on a scale from 0 - 100, where lower scores represented better functional status.
Time Frame: Baseline (1 week), Mid-Treatment (2 weeks post-baseline), Post-Treatment (4 weeks post-baseline)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Light Therapy A (Bright) Via the Re-Timer® | Light Therapy B (Dim) Via the Re-Timer®
Number analyzed (Participants) | 29 | 28
score on a scale
  Baseline (1 week) | 40.8 (13.2) | 45.3 (19.0)
  Mid-Treatment (completed 2 Weeks following baseline) | 38.0 (13.5) | 39.4 (18.3)
  Post Treatment (completed 4 Weeks following baseline) | 32.2 (12.3) | 32.7 (19.2)
Statistical Analysis 1: Comparison: Light Therapy A (Bright) Via the Re-Timer® vs Light Therapy B (Dim) Via the Re-Timer®; Test of between-arm difference at mid-treatment; Test type: Superiority; p = 0.28, Mixed Models Analysis; The comparison was done using a mixed model with assessments at 3 time points (pre-treatment, mid-treatment, and end of treatment); Mean Difference (Net) = 3.80, 95% CI 2-sided [-3.03 to 10.64], Standard Error of Mean 3.49
Statistical Analysis 2: Comparison: Light Therapy A (Bright) Via the Re-Timer® vs Light Therapy B (Dim) Via the Re-Timer®; Test of between-arm difference at end of treatment; Test type: Superiority; p = 0.21, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = 4.48, 95% CI 2-sided [-2.44 to 11.40], Standard Error of Mean 3.53

2. Secondary Outcome: Heat Pain Threshold Assessed by the Heat Pain Sensitivity Test
Description: Pain threshold was assessed during a heat pain sensitivity task using a Medoc TSAII NeuroSensory Analyzer and an ascending method of limits protocol. The threshold was the temperature (in degrees Celsius) at which the participant reported the stimulus felt painful.
Time Frame: Baseline (1 week), Mid-Treatment (2 weeks post-baseline), Post-Treatment (4 weeks post-baseline)
Population: Due to COVID-19's impact on in-person visits, close, in-person measurements were stopped. Only earlier participants' data is available.
Measure: Mean (Standard Deviation); unit: Degrees Celsius
Arm/Group | Light Therapy A (Bright) Via the Re-Timer® | Light Therapy B (Dim) Via the Re-Timer®
Number analyzed (Participants) | 16 | 14
Degrees Celsius
  Baseline (1 week) | 41.9 (3.3) | 41.9 (3.4)
  Mid-Treatment (completed 2 weeks post-baseline) | 42.4 (3.5) | 41.8 (3.1)
  Post-Treatment (completed 4 weeks post-baseline) | 42.7 (3.1) | 42.6 (3.3)

3. Secondary Outcome: Heat Pain Tolerance Assessed by the Heat Pain Sensitivity Test
Description: Pain tolerance was assessed during a heat pain sensitivity task using a Medoc TSAII NeuroSensory Analyzer and an ascending method of limits protocol. The tolerance was the temperature (in degrees Celsius) at which the participant reported the stimulus was so painful that they had to stop.
Time Frame: Baseline (1 week), Mid-Treatment (2 weeks post-baseline), Post-Treatment (4 weeks post-baseline).
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Degrees Celsius
Arm/Group | Light Therapy A (Bright) Via the Re-Timer® | Light Therapy B (Dim) Via the Re-Timer®
Number analyzed (Participants) | 16 | 14
Degrees Celsius
  Baseline (1 week) | 47.6 (1.8) | 46.2 (2.2)
  Mid-Treatment (completed 2 weeks post-baseline) | 47.9 (1.6) | 46.2 (2.0)
  Post-Treatment (completed 4 weeks post-baseline) | 47.8 (1.5) | 46.8 (2.0)

4. Secondary Outcome: Patient Reported Outcomes Measurement Information System (PROMIS) Pain Intensity Score
Description: Pain was assessed with the Patient-Reported Outcomes Measurement Information System (PROMIS) Pain Intensity 3a short form, which assesses worst and average pain in the past 7 days (1=no pain to 5=very severe) and current level of pain (1=no pain to 5= very severe). Scores were summed and converted to a T score metric (mean ±SD, 50 ±10); higher scores indicate more pain.
Time Frame: Baseline (1 week), Mid-Treatment (2 weeks post-baseline), Post-Treatment (4 weeks post-baseline).
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Light Therapy A (Bright) Via the Re-Timer® | Light Therapy B (Dim) Via the Re-Timer®
Number analyzed (Participants) | 29 | 28
T-score
  Baseline (1 week) | 51.0 (5.6) | 51.6 (5.4)
  Mid-Treatment (completed 2 weeks post-baseline) | 49.8 (5.5) | 50.4 (5.8)
  Post-Treatment (completed 4 weeks post-baseline) | 47.9 (4.4) | 49.6 (6.2)

ADVERSE EVENTS:
Time Frame: Through study completion, an average of 5 weeks.
Description: Systematic Assessment for Treatment Emergent Events (SAFTEE) Questionnaire, a self-reported measure of physical and emotional symptoms experienced in the past week.
Arm/Group | Light Therapy A (Bright) Via the Re-Timer® | Light Therapy B (Dim) Via the Re-Timer®
All-Cause Mortality (participants affected / at risk) | 0/29 | 0/28
Serious Adverse Events (participants affected / at risk) | 0/29 | 0/28
Other Adverse Events (participants affected / at risk) | 0/29 | 0/28

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-02-22): https://cdn.clinicaltrials.gov/large-docs/08/NCT03794908/Prot_SAP_001.pdf
  • Informed Consent Form (2021-01-21): https://cdn.clinicaltrials.gov/large-docs/08/NCT03794908/ICF_000.pdf